CLINICAL TRIAL: NCT02599480
Title: A Multi-centre Randomized, Placebo-controlled Trial of Mirabegron, a New beta3-adrenergic Receptor Agonist on Left Ventricular Mass and Diastolic Function in Patients With Structural Heart Disease
Brief Title: Assessment of Efficacy of Mirabegron, a New beta3-adrenergic Receptor in the Prevention of Heart Failure
Acronym: Beta3_LVH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jean-Luc Balligand (Other)
Collaborators: Zentrum für Klinische Studien Leipzig (Other); European Clinical Research Infrastructure Network (Other); European Society of Cardiology (Network); European Commission (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Northern Lisbon Hospital Center (Other); University of Athens (Other); Center for Cardiovascular Research Berlin (Other); Wroclaw Medical University (Other); Papa Giovanni XXIII Hospital (Other); Nantes University Hospital (Other); University Medical Center Goettingen (Other); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Jean-Luc Balligand, Professor, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beta3_LVH V1.0
Record Dates: First submitted 2015-10-30; First posted 2015-11-06 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hypertrophy, Left Ventricular
Keywords: HFpEF; left ventricular hypertrophy; cardiac remodeling,
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — mirabegron; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mirabegron (Active Comparator): Patients will be orally administererd with 50 mg of mirabegron once a day during 12 months.
  Interventions: Drug: mirabegron; Procedure: Echocardiography; Procedure: Cardiac MRI; Procedure: Maximal exercise capacity; Procedure: Blood sampling; Procedure: Endothelial function measurement; Radiation: 18FDG-PET
- Placebo (Placebo Comparator): Patients will be orally administererd with a placebo once a day during 12 months.
  Interventions: Procedure: Echocardiography; Procedure: Cardiac MRI; Procedure: Maximal exercise capacity; Procedure: Blood sampling; Procedure: Endothelial function measurement; Radiation: 18FDG-PET

INTERVENTIONS:
Drug: mirabegron — 50 mg daily during 12 months
  Other Names: Betmiga, Myrbetriq
  Arms: mirabegron
Procedure: Echocardiography — Echocardiography
Procedure: Cardiac MRI — Cardiac MRI
Procedure: Maximal exercise capacity — Maximal exercise capacity
Procedure: Blood sampling — Blood sampling for study assessments and future exploratory studies.
Procedure: Endothelial function measurement — EndoPAT assessment
Radiation: 18FDG-PET — PET scanning for beige/brown fat activation

SUMMARY:
This study will assess the efficacy of mirabegron, a new beta3-adrenergic receptor in the prevention of heart failure. This is a two armed, prospective, randomized, placebo-controlled, multi-centric european phase IIb trial with placebo and mirabegron distributed in a 1:1 fashion. The patients enrolled will have cardiac structural remodeling with or without symptoms of heart failure (maximum NYHA II).

Patients will be monitored for change in left ventricular mass (assessed by cardiac MRI) and/or changes in diastolic function (assessed by echocardiography) after 12 months of treatment.

DETAILED DESCRIPTION:
Background Heart failure (HF) represents a major and growing public health burden. Patients with HF are classically divided into two groups: those with HF with preserved ejection fraction (HFpEF), and those with HF and reduced ejection fraction (HFrEF). As HF is a progressive disorder increasing with age, the proportion of these patients is rising due to the aging of the population. Beside costs, HFpEF also puts a heavy burden on the quality of life of (mostly elderly) patients, with a loss of autonomy and the dyscomfort of repeated hospitalisations. Therefore, HFpEF is a chronic, costly, debilitating disease.

A major contributor to HFpEF is myocardial remodelling, e.g. hypertrophy and fibrosis, as well as cellular functional/structural modifications leading to alteration in contractile properties and ventricular distensibility. Unfortunately, there are currently no evidence-based treatment strategies.

Study claim The proposed clinical trial will provide a proof of concept in humans for the clinical efficacy of a novel therapeutic concept: β3AR activation to attenuate/prevent cardiac remodeling. Recently, a new, specific agonist at human β3-AR (mirabegron) with higher benefit/risk balance was developed and marketed for clinical use in a non-cardiovascular disease (overactive bladder disease). The trial will test the drug repurposing of mirabegron for the prevention of cardiac remodeling leading to HFpEF.

Using pre-clinical models, the investigators demonstrated that activation of β3AR attenuates myocardial hypertrophy and fibrosis in response to neurohormonal or hemodynamic stresses, without compromising LV function. Therefore, the recent availability of this new drug offers the possibility to test the potential benefit of mirabegron (vs placebo) as add-on therapy (on top of standard care) to prevent/delay myocardial remodelling in patients at high risk of developing HFpEF.

Who can participate? Patients with structural cardiac disease with or without HF symptoms (max. NYHA 2).

What does the study involve? Patients will be requested to go 5 times to the hospital to perform cardiac MRI (3X), echocardiography (3X), exercise tolerance test (2X), Pet scanning (2X) and blood sampling (4X).

Who is the sponsor? The Université catholique de Louvain (UCL) is the academic sponsor and Prof. Jean-Luc Balligand is the principal coordinator of the study.

Who is funding the study? Beta3_LVH is an investigator-initiated project funded by a Horizon 2020 grant from the European Commission.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Arterial hypertension on stable therapy according to current guideline algorithms (including stable medication for at least four weeks before inclusion),
* Morphological signs of structural cardiac remodelling by echocardiography, i.e. increased LV mass index (110 g/m2 or higher for female; 134 g/m2 or higher for male subjects (Devereux, Reichek 1977)) or end-diastolic wall thickness > or equal to 13 mm in at least one wall segment
* Patients may have atrial fibrillation (AF), but with well-regulated ventricular response, i.e. heart rate<100/min (RACE II - (Groenveld et al. 2013, 2013)),
* Written informed consent
* For subjects unable to read and/or write, oral informed consent observed by an independent witness is acceptable if the subject has fully understood oral information given by the Investigator. The witness should sign the consent form on behalf of the subject.

Exclusion Criteria:

* Unstable hypertension with systolic BP≥160 mm Hg and/or diastolic BP≥100 mm Hg (based on office measurement, not ambulatory measurement)
* Documented ischemic cardiac disease
* History of hospitalization for overt heart failure within last 12 months
* Patients after heart transplantation
* Genetic hypertrophic or dilated cardiomyopathy
* Dysthyroidism.
* Severe valvulopathy
* NYHA-class > II
* BMI >40 kg/m2
* EF < 50%, regardless of symptoms
* Known other cause (i.e. COPD) of respiratory dysfunction; patients under positive pressure (CPAP) treatment for sleep apnea syndrome may be included, provided they have been under regular treatment for at least one year before inclusion in the study
* eGFR < 30 ml/min (by MDRD formula)
* Abnormal liver function tests
* Type I diabetes, complicated type II diabetes
* Patients with anemia
* Patients with bladder outlet obstruction
* Patients using antimuscarinic cholinergic drugs for treatment of OAB
* Current use of digitalis, bupranolol, propranolol, nebivolol
* Patients continuously treated with Sildenafil or other PDE5 inhibitors.
* Current use of antifungal azole derivatives (fluconazole, itraconazole, miconazole, posaconazole, voriconazole)
* Current treatment with mirabegron or indication for future treatment with mirabegron due to other indications
* Contraindication for MRI
* Pregnant or nursing women
* Participation in any other interventional trial
* Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (hormonal implant, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial (participants using a hormone-based method have to be informed of possible effects from the trial medication on contraception)
* Contraindication to mirabegron (e.g. hypersensitivity) or any other components of the trial medication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass index (LVMI) | 12 months
  Change in left ventricular mass index (LVMI in g/m2, defined as left ventricular mass divided by body surface) measured at baseline and 12 months after randomisation.
Change in diastolic function | 12 months
  Change in diastolic function, assessed as the ratio of peak early transmitral ventricular filling velocity to early diastolic tissue Doppler velocity (E/e') measured at baseline and 12 months after randomisation.

SECONDARY OUTCOMES:
Cardiac fibrosis | 12 months
  Cardiac fibrosis at baseline and at 12 months. Fibrosis is a key pathogenic mechanism of diastolic dysfunction, which is at the origin of HFpEF
Left atrial volume index | 12 months
  Left atrial volume index at baseline and at 12 months. This parameter determines diastolic filling (and was shown to predict treatment efficacy in HFpEF in the J-DHF trial (Yamamoto et al. 2013))
LV mass index (by cardiac MRI) | 6 months
  LV mass index (by cardiac MRI) at 6 months,
Diastolic function (E/e') | 6 months
  Diastolic function (E/e') at 6 months
serum biomarkers | 3, 6, 12 months
  serum biomarkers (Galectin3, GDF15, NT-proBNP, hsTnT)
metabolic parameters | 3, 6, 12 months
  metabolic parameters (fasting glucose, modified HOMA test, HbA1c, serum lipids)
Maximal exercise capacity | 12 months
  Maximal exercise capacity (peak VO2) at baseline and 12 months.
Emergence of treatment-related adverse events | 12 months
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Balligand, Prof. MD, Principal Investigator — Université Catholique de Louvain
Locations (10):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Nantes university hospital (CHU Nantes), Nantes, France
- Germany (3):
  - Center for Cardiovascular Research Berlin (CCR/Charité), Berlin
  - University Medical Center Göttingen (UMG-GOE), Göttingen
  - University of Leipzig, Leipzig
- Athens University Medical School (NKUA), Athens, Greece
- Hospital "Papa Giovanni XXIII" (HPG23), Bergamo, Italy
- Department of Heart Diseases at Wroclaw Medical University (UMW), Wroclaw, Poland
- Association for Research and Development of the Faculty of Medicine (AIDFM), Lisbon, Portugal
- University of Oxford - Division of Cardiovascular Medicine (UOXF), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data required to reach aims in an approved proposal, after de-identification, will be made available to investigators whose proposed use of the data has been approved by the study's Executive Committee. Proposals may be submitted up to 36 months after publication of the study results and should be directed to Jean-Luc.Balligand@uclouvain.be.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: up to 36 months after publication of the study results
Access Criteria: Upon approval by the study Steering Committee of a valid proposal by requesters

REFERENCES:
- [Background] Belge C, Hammond J, Dubois-Deruy E, Manoury B, Hamelet J, Beauloye C, Markl A, Pouleur AC, Bertrand L, Esfahani H, Jnaoui K, Gotz KR, Nikolaev VO, Vanderper A, Herijgers P, Lobysheva I, Iaccarino G, Hilfiker-Kleiner D, Tavernier G, Langin D, Dessy C, Balligand JL. Enhanced expression of beta3-adrenoceptors in cardiac myocytes attenuates neurohormone-induced hypertrophic remodeling through nitric oxide synthase. Circulation. 2014 Jan 28;129(4):451-62. doi: 10.1161/CIRCULATIONAHA.113.004940. Epub 2013 Nov 4. PMID 24190960
- [Background] Balligand JL. beta(3)-Adrenoceptor stimulation on top of beta(1)-adrenoceptor blockade "Stop or Encore?". J Am Coll Cardiol. 2009 Apr 28;53(17):1539-42. doi: 10.1016/j.jacc.2009.01.048. No abstract available. PMID 19389565
- [Background] Dessy C, Balligand JL. Beta3-adrenergic receptors in cardiac and vascular tissues emerging concepts and therapeutic perspectives. Adv Pharmacol. 2010;59:135-63. doi: 10.1016/S1054-3589(10)59005-7. PMID 20933201
- [Derived] Menghoum N, Badii MC, Leroy M, Parra M, Roy C, Lejeune S, Vancraeynest D, Pasquet A, Brito D, Casadei B, Depoix C, Filippatos G, Gruson D, Edelmann F, Ferreira VM, Lhommel R, Mahmod M, Neubauer S, Persu A, Piechnik S, Hellenkamp K, Ikonomidis I, Krakowiak B, Pieske B, Pieske-Kraigher E, Pinto F, Ponikowski P, Senni M, Trochu JN, Van Overstraeten N, Wachter R, Gerber BL, Balligand JL, Beauloye C, Pouleur AC. Exploring the impact of metabolic comorbidities on epicardial adipose tissue in heart failure with preserved ejection fraction. Cardiovasc Diabetol. 2025 Mar 22;24(1):134. doi: 10.1186/s12933-025-02688-7. PMID 40121452
- [Derived] Balligand JL, Brito D, Brosteanu O, Casadei B, Depoix C, Edelmann F, Ferreira V, Filippatos G, Gerber B, Gruson D, Hasenclever D, Hellenkamp K, Ikonomidis I, Krakowiak B, Lhommel R, Mahmod M, Neubauer S, Persu A, Piechnik S, Pieske B, Pieske-Kraigher E, Pinto F, Ponikowski P, Senni M, Trochu JN, Van Overstraeten N, Wachter R, Pouleur AC. Repurposing the beta3-Adrenergic Receptor Agonist Mirabegron in Patients With Structural Cardiac Disease: The Beta3-LVH Phase 2b Randomized Clinical Trial. JAMA Cardiol. 2023 Nov 1;8(11):1031-1040. doi: 10.1001/jamacardio.2023.3003. PMID 37728907

DOCUMENTS (3):
  • Study Protocol (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT02599480/Prot_000.pdf
  • Statistical Analysis Plan: Planned analyses (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02599480/SAP_001.pdf
  • Statistical Analysis Plan: Trial results according to ICH E3 (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT02599480/SAP_002.pdf